CLINICAL TRIAL: NCT00826969
Title: Ciclesonide for the Treatment of Airway Hyperresponsiveness. The Mannitol-Asthma-Ciclesonide Study (MACS). A Double-blind, Randomized, Parallel Group Study.
Brief Title: Ciclesonide for the Treatment of Airway Hyperresponsiveness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/CH-101; U1111-1137-3949 (Registry Identifier: WHO)
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide
MeSH Terms: conditions — Asthma | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Ciclesonide 320µg
  Interventions: Drug: Ciclesonide
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclesonide — 320µg Ciclesonide versus Placebo
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The study objective is to investigate in a placebo-controlled, double-blind manner the effect of inhaled corticosteroid (ciclesonide) on airway hyperresponsiveness measured as having PD15 mannitol. Treatment medication will be administered as follows: 320 microgram ciclesonide or placebo will be inhaled once daily. The study duration consists of a treatment period of 4 weeks. The study will provide further data on safety of ciclesonide.

ELIGIBILITY:
Inclusion Criteria:

1. Referred to the pulmonology department of the university hospital Basel because of suspected asthma defined as respiratory symptoms like wheezing or cough or chest tightness.
2. Asthma symptoms partly controlled according to GINA (October 2006) 1 week prior to randomization
3. FEV1 ≥ 70% predicted
4. 18 - 70 years old

Exclusion Criteria:

1. Smoker and ex-smoker with >10 pack years
2. COPD
3. Upper respiratory tract infection within the past 4 weeks.
4. ICS or oral steroids during the previous month before inclusion
5. b-blockers within the past 4 weeks
6. Current treatment with medication as defined in section concomitant medication (ICS other than study medication, ß-blockers)
7. Pregnancy
8. Known malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-09; Primary Completion 2010-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change of hyper-responsiveness to mannitol assessed by PD15FEV1 after 4 weeks of treatment with ciclesonide vs Placebo | 4 weeks

SECONDARY OUTCOMES:
RDR mannitol (response-dose-ratio = %fall in FEV1 / provocation dose given) | 4 weeks
Responsiveness to methacholine (PD20FEV1 ) and RDR methacholine after 4 weeks of treatment | 4 weeks
Level of exhaled nitric oxide after 4 weeks of treatment | 4 weeks
mean improvement of FEV1 and PEF, mean change of the asthma control questionnaire ACQ (Juniper) | 4 weeks
Mean change of ACQ after 4 weeks of treatment | 4 weeks
Mean change of AQLQ after 4 weeks of treatment | 4 weeks
Mean change of symptoms, rescue medication use, nocturnal awakening according to GINA after 4 weeks of treatment | 4 weeks
Exacerbation rates during the 4 weeks of treatment | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Nycomed, Basel, Switzerland

REFERENCES:
- See also: BY9010-CH-101-RDS-2012-10-29.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4509&filename=BY9010-CH-101-RDS-2012-10-29.pdf